CLINICAL TRIAL: NCT06463483
Title: Glucose Control With Medtronic 780G System in Adults With Diabetes and Advanced Renal Disease
Brief Title: Automated Insulin Delivery in Adults With Advanced Kidney Disease
Acronym: AIDkidney
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24HH8885
Record Dates: First submitted 2024-06-10; First posted 2024-06-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus
Keywords: Diabetes; Automated Insulin Delivery; Dialysis; Chronic Kidney Diseases; Insulin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Insulin Resistance | interventions — Drug Delivery Systems; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Automated insulin delivery using Medtronic 780G System (Experimental)
  Interventions: Device: Medtronic 780G System
- Usual care plus continuous glucose monitoring (Other)
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Medtronic 780G System — Automated insulin delivery using Medtronic 780G system
  Arms: Automated insulin delivery using Medtronic 780G System
Device: Continuous Glucose Monitoring — Usual care with continuous glucose monitoring
  Arms: Usual care plus continuous glucose monitoring

SUMMARY:
Diabetes is the leading cause of kidney failure in the UK. Many people with diabetes and advanced kidney failure inject themselves with insulin and do finger-prick blood glucose tests. Managing diabetes in people with advanced kidney disease is hard, with fluctuating glucose levels and an increased risk of unsafe low glucose levels.

There are currently continuous glucose monitors (CGM), which allow people to monitor glucose without painful fingerprick tests. CGM can be combined with insulin pumps to create automated insulin delivery systems (AID) that deliver insulin automatically to control glucose. AID systems are currently used in people with type 1 diabetes, but they are not used in people with type 2 diabetes. There is little information on how these systems might help people with diabetes and advanced kidney failure and on dialysis.

This study will investigate whether automated insulin delivery can improve glucose levels and quality of life in people with diabetes treated with more than one insulin injection with advanced kidney failure and/or undergoing regular dialysis treatment. This study will be a feasibility study conducted in a single centre (Imperial College, London) and be of a cross-over design. The study will aim to complete 12 people. Participants will wear a glucose sensor at the start. In random order, half will start AID followed by the usual treatment, while the other half will start the usual treatment followed by AID treatment. The duration of each treatment stage is eight weeks. The study will last about 22 weeks for each participant. Investigators will compare the glucose levels in the AID group with the usual care group to see if there is a difference. Questionnaires and interviews will help us understand participants' experiences. Investigators will carefully monitor the safety of participants.

DETAILED DESCRIPTION:
This will be a single-centre, prospective, open-label, two-stage, randomized crossover study comparing automated subcutaneous insulin delivery (AID), also known as Hybrid Closed Loop (HCL) therapy using the 780G system with usual insulin therapy plus continuous glucose monitoring (CGM) in people with type 1 and type 2 diabetes complicated by advanced renal disease and managed with insulin. The study will be conducted at Imperial College Healthcare NHS Trust.

Duration of each treatment arm is 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-70 years inclusive
* 2. Type 1 diabetes of at least 1-year duration or insulin-requiring type 2 diabetes managed with multiple daily injections (MDI [ie separate rapid-acting and basal insulin injections]) or insulin pump therapy (CSII)
* 3. The HbA1c <10.5% (<91 mmol/mol)
* 4. The total daily dose of insulin <200Units
* 5. The participant is willing and able to implement the study requirements.
* 6. Participant has advanced renal disease (Group A: Stage 3b or greater renal failure (eGFR <45millilitres/minute/1.73m2); Group B: ESKD requiring peritoneal dialysis; Group C: ESKD requiring haemodialysis
* 7. Participants (and carer where applicable) should be able to speak and understand English sufficiently for safe study conduct
* 8. The participant has internet or smartphone access, enabling upload of the 780G system data to cloud-based software

Exclusion Criteria:

* 1. The participant is already using an AID system
* 2. The participant is treated with sulphonylureas (SGLT2 inhibitors, metformin, and GLP1 analogues may be used within regulatory guidelines) in pre-dialysis participants (Group A). In Groups B & C, noninsulin glucose-lowering therapies are not permitted, with the exception of GLP1 agonists used in preparation for transplantation
* 3. The participant has a recent history of diabetic ketoacidosis (<6 months)
* 4. The use of systemic steroid therapy within the past four weeks (stable doses of steroids for >8 weeks permitted)
* 5. The participant has significant cognitive impairment or major psychiatric history affecting safe study conduct
* 6. Known significant allergy to tape/ adhesives
* 7. Women who are pregnant or planning pregnancy
* 8. The participant has an active major life-threatening illness limiting the participants life expectancy to <6 months
* 9. The participant is on hydroxyurea treatment or taking regular / daily paracetamol treatment (sensor interference)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Percent time in sensor glucose target range (3.9-10.0 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (3.9-10.0 mmol/L) with Automated Insulin Delivery (AID) versus Usual Care measured during the final 3 weeks of each study stage.

SECONDARY OUTCOMES:
Percent time in sensor glucose target range (<3.0 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<3.0 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (<3.9 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<3.9 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (>10 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<10 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (<2.8 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<2.8 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (<3.3 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<3.3 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (>13.9 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<13.9 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (>16.7 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (<16.7 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Percent time in sensor glucose target range (3.9-7.8 mmol/L) | 3 weeks
  Percent time in sensor glucose target range (3.9-7.8 mmol/L) with AID versus Usual Care, measured during the final 3 weeks of each study stage
Mean sensor glucose | 3 weeks
  Mean sensor glucose with AID versus Usual Care, measured during the final 3 weeks of each study stage
Standard deviation and coefficient of variation of sensor glucose | 3 weeks
  Standard deviation and coefficient of variation of sensor glucose with AID versus Usual Care, measured during the final 3 weeks of each study stage
The Diabetes Treatment Satisfaction Questionnaire status | 8 weeks
  The Diabetes Treatment Satisfaction Questionnaire status with AID versus Usual Care
Hypoglycaemia Fear Survey | 8 weeks
  Hypoglycaemia Fear Survey with AID versus Usual Care
EQ-5D-5L | 8 weeks
  EQ-5D-5L with AID versus Usual Care
Episodes of CGM time in <3.0mmol/L range lasting >15minutes | 3 weeks
  Episodes of CGM time in <3.0mmol/L range lasting >15minutes with AID versus Usual Care
Number of hospital admissions with diabetic ketoacidosis or hyperosmolar non-ketotic hyperglycaemia | 8 weeks
  Number of hospital admissions with diabetic ketoacidosis or hyperosmolar non-ketotic hyperglycaemia with AID versus Usual Care
Number of hospitalised and non-hospitalised patients with severe hypoglycaemia | 8 weeks
  Number of hospitalised and non-hospitalised patients with severe hypoglycaemia with AID versus Usual Care

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Background] Boughton CK, Tripyla A, Hartnell S, Daly A, Herzig D, Wilinska ME, Czerlau C, Fry A, Bally L, Hovorka R. Fully automated closed-loop glucose control compared with standard insulin therapy in adults with type 2 diabetes requiring dialysis: an open-label, randomized crossover trial. Nat Med. 2021 Aug;27(8):1471-1476. doi: 10.1038/s41591-021-01453-z. Epub 2021 Aug 4. PMID 34349267
- [Background] Bally L, Gubler P, Thabit H, Hartnell S, Ruan Y, Wilinska ME, Evans ML, Semmo M, Vogt B, Coll AP, Stettler C, Hovorka R. Fully closed-loop insulin delivery improves glucose control of inpatients with type 2 diabetes receiving hemodialysis. Kidney Int. 2019 Sep;96(3):593-596. doi: 10.1016/j.kint.2019.03.006. Epub 2019 Mar 20. PMID 31133457
- [Background] Lu JC, Lee P, Ierino F, MacIsaac RJ, Ekinci E, O'Neal D. Challenges of Glycemic Control in People With Diabetes and Advanced Kidney Disease and the Potential of Automated Insulin Delivery. J Diabetes Sci Technol. 2024 Nov;18(6):1500-1508. doi: 10.1177/19322968231174040. Epub 2023 May 10. PMID 37162092